CLINICAL TRIAL: NCT04723576
Title: Mental and Physical Well-Being of Frontline Health Care Workers During Coronavirus Disease 2019 (COVID-19)
Acronym: COVER-HCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Stanford University (Other); Clinical Directors Network (Network); Vizient (Unknown)
Responsible Party: Principal Investigator, Lisa Meredith, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COVID-2020C2-10721; COVID-2020C2-10721 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2021-01-14; First posted 2021-01-25 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: healthcare worker; stress; fatigue; anxiety; burnout; COVID-19; stress first aid
MeSH Terms: conditions — Fatigue; Anxiety Disorders; Burnout, Psychological; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking of research staff will be performed to the extent possible in this study. The survey data can be analyzed in a blinded fashion. However, due to the nature of qualitative research (described below), masking will not be possible for this data collection effort. Given that no qualitative research can be performed in a blinded way, we do not anticipate the lack of masking to affect our qualitative results adversely.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress First Aid (Experimental): The cluster Randomized Controlled Trial (cRCT) will be comprised of three cohorts of matched pairs representing approximately 40 diverse sites (12-15 pairs of hospitals hospitals and 5-7 pairs of clinics/practices) to determine whether SFA for frontline HCWs improves mental and physical well-being compared to Usual Care (UC). Each pair will be assigned to either SFA or UC using a simple 1:1 randomization. SFA sites will implement SFA through a "train-the-trainer" model.
  Interventions: Behavioral: Stress First Aid
- Usual Care (No Intervention): The cRCT will be comprised of three cohorts of matched pairs representing approximately 40 diverse sites (12-15 pairs of hospitals hospitals and 5-7 pairs of clinics/practices) to determine whether SFA for frontline HCWs improves mental and physical well-being compared to Usual Care (UC). Each pair will be assigned to either SFA or UC using a simple 1:1 randomization. UC sites will not implement SFA during the study period but will be given full access to all implementation materials following the conclusion of their participation.

INTERVENTIONS:
Behavioral: Stress First Aid — Stress First Aid (SFA) is an evidence-based intervention to mitigate the psychosocial impact of COVID-19 on Health Care Workers (HCWs). SFA was initially developed for the United States Navy and Marine Corps as a framework of actions for peer support delivered by individuals without mental health training. SFA is designed to teach simple, supportive actions that can be seamlessly integrated into work environments. SFA training focuses on five essential principles: cover (restore and support a sense of safety), calm (encourage simple strategies such as breathing), connect (engage in and promote social support), competence (improve ability to address crucial needs and concerns), and confidence (increase hope and limit self-doubt and guilt). In this study, we are adapting the SFA model to include HCW-specific examples of SFA actions and case scenarios specific to the COVID-19 pandemic and will implement SFA using a "train-the trainer" model.
  Arms: Stress First Aid

SUMMARY:
Study to support the mental and physical well-being of US health care workers during the COVID-19 pandemic and ensure high-quality care for patients through Stress First Aid.

DETAILED DESCRIPTION:
The goal of the project is to support the mental and physical well-being of U.S. health care workers (HCWs) during the COVID-19 pandemic to ensure high-quality care for patients, by establishing the effectiveness of a tailored Stress First Aid (SFA) intervention, compared to usual care (UC). The RAND Corporation will conduct a cluster randomized controlled trial (cRCT) with three cohorts containing matched pairs in approximately 40 diverse sites (hospitals and clinics) to evaluate whether SFA for HCWs improves mental and physical well-being compared to UC. Sequential roll-out of the intervention to three cohorts will allow investigators to quickly incorporate lessons learned and stakeholder feedback from each iteration into subsequent trainings, and share actionable findings given the urgency due to the pandemic. The end result will be an SFA toolkit tailored for HCWs that can be implemented and scaleable across multiple settings. The proposed SFA intervention addresses an important and compelling clinical care delivery challenge during COVID-19 by improving the mental well-being of HCWs, who will benefit directly and be better equipped to provide higher quality, more sustained, and more patient-centered care to patients. The specific aims of the project are to: (1) test the comparative effectiveness of SFA versus UC on mental and physical well-being (quantitative); (2) understand and document any UC activities to support HCW well-being prior to implementing SFA across sites; and (3) assess the experiences of HCWs and sites with SFA (acceptability, likelihood of uptake, lessons learned) and impact on HCW well-being (qualitative).

ELIGIBILITY:
Inclusion Criteria:

* Health care workers and patient-facing support staff (e.g., front desk staff)

Exclusion Criteria:

* Non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7444 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Renzi, Study Director — RAND
Locations (2):
- United States (2):
  - Clinical Directors Network, Inc, New York, New York
  - Vizient Inc., Irving, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will follow the funder's protocol for uploading data.
Supporting Information: Study Protocol, ICF
Time Frame: December 2022
Access Criteria: The study data are available to qualified researchers and provided a de-identified copy of the study data and related documentation to the REGENTS OF THE UNIVERSITY OF MICHIGAN on behalf of the INTER-UNIVERSITY CONSORTIUM FOR POLITICAL AND SOCIAL RESEARCH (ICPSR) for the purpose of allowing ICPSR to examine, process, and distribute the data to qualified researchers as determined by ICPSR.
URL: http://www.cdc.gov/nchs/data/nchs_microdata_release_policy_4-02A.pdf

REFERENCES:
- [Background] Dong L, Meredith LS, Farmer CM, Ahluwalia SC, Chen PG, Bouskill K, Han B, Qureshi N, Dalton S, Watson P, Schnurr PP, Davis K, Tobin JN, Cassells A, Gidengil CA. Protecting the mental and physical well-being of frontline health care workers during COVID-19: Study protocol of a cluster randomized controlled trial. Contemp Clin Trials. 2022 Jun;117:106768. doi: 10.1016/j.cct.2022.106768. Epub 2022 Apr 22. PMID 35470104
- [Background] Meredith LS, Ahluwalia S, Chen PG, Dong L, Farmer CM, Bouskill KE, Dalton S, Qureshi N, Blagg T, Timmins G, Schulson LB, Huilgol SS, Han B, Williamson S, Watson P, Schnurr PP, Martineau M, Davis K, Cassells A, Tobin JN, Gidengil C. Testing an Intervention to Improve Health Care Worker Well-Being During the COVID-19 Pandemic: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e244192. doi: 10.1001/jamanetworkopen.2024.4192. PMID 38687482
- [Background] Bandini JI, Ahluwalia SC, Timmins G, Bialas A, Meredith L, Gidengil C. "It Haunts Me": Impact of COVID-19 Deaths on Frontline Clinicians In Acute Care Settings-A Qualitative Study. Am J Crit Care. 2023 Sep 1;32(5):368-374. doi: 10.4037/ajcc2023257. PMID 37652873
- [Background] Timmins GT, Bandini JI, Ahluwalia SC, Bialas A, Meredith LS, Gidengil C. 'You just don't feel like your work goes recognised': healthcare worker experiences of tension related to public discourse around the COVID-19 pandemic. BMJ Lead. 2024 Dec 23;8(4):324-328. doi: 10.1136/leader-2024-000983. PMID 38553036
- [Background] Qureshi N, Huilgol SS, Timmins G, Meredith LS, Gidengil CA. Misaligned Supports: Differences in Reported Health Care Worker Well-being Supports Provided and Needed During the COVID-19 Pandemic. Am J Health Promot. 2025 Jan;39(1):63-75. doi: 10.1177/08901171241255764. Epub 2024 Jun 21. PMID 38907369
- [Derived] Timmins G, Williamson S, Cassells A, Davis K, Dong L, Tobin JN, Gidengil C, Meredith LS, Chen PG. Health care worker experiences with a brief peer support and well-being intervention during the COVID-19 pandemic. BMC Health Serv Res. 2025 Sep 30;25(1):1253. doi: 10.1186/s12913-025-13268-6. PMID 41029307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 hospitals and Federally Qualified Health Centers (FQHCs) throughout the US were recruited in 3 consecutive cohorts and enrolled from March 2021 through July 2022. Participating sites were matched as pairs by type, size, and COVID-19 burden and then randomized to the intervention arm or usual care arm.
Pre-assignment Details: Health care worker (HCW) participants completed a pre-intervention survey prior to randomization.
Units Other Than Participants: FQHCs/Hospitals
Groups:
- Stress First Aid: The cRCT will be comprised of three cohorts of matched pairs representing approximately 40 diverse sites (12-15 pairs of hospitals hospitals and 5-7 pairs of clinics/practices) to determine whether SFA for frontline HCWs improves mental and physical well-being compared to Usual Care (UC). Each pair will be assigned to either SFA or UC using a simple 1:1 randomization. SFA sites will implement SFA through a "train-the-trainer" model.
  Stress First Aid: Stress First Aid (SFA) is an evidence-based intervention to mitigate the psychosocial impact of COVID-19 on Health Care Workers (HCWs). SFA was initially developed for the United States Navy and Marine Corps as a framework of actions for peer support delivered by individuals without mental health training. SFA is designed to teach simple, supportive actions that can be seamlessly integrated into work environments. SFA training focuses on five essential principles: cover (restore and support a sense of safety), calm (encourage simple strategies such as breathing), connect (engage in and promote social support), competence (improve ability to address crucial needs and concerns), and confidence (increase hope and limit self-doubt and guilt). In this study, we are adapting the SFA model to include HCW-specific examples of SFA actions and case scenarios specific to the COVID-19 pandemic and will implement SFA using a "train-the trainer" model.
Period: Overall Study
Arm/Group | Stress First Aid | Usual Care
Started | 2995; 14 FQHCs/Hospitals | 4449; 14 FQHCs/Hospitals
Completed | 862; 14 FQHCs/Hospitals | 1215; 14 FQHCs/Hospitals
Not Completed | 2133; 0 FQHCs/Hospitals | 3234; 0 FQHCs/Hospitals
Not completed — Withdrawal by Subject | 2133 | 3234

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stress First Aid | Usual Care | Total
Number analyzed (Participants) | 862 | 1215 | 2077
Age, Customized [Count of Participants; unit: Participants]
  <= 30 | 223 | 275 | 498
  31-50 | 486 | 696 | 1182
  >= 51 | 152 | 240 | 392
  Missing | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Numbers differ due to missing responses.
  Participants
    number analyzed (Participants) | 855 | 1206 | 2061
    Female | 696 | 947 | 1643
    Male | 159 | 259 | 418
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 132 | 145 | 277
  Hispanic or Latino//Latina | 157 | 259 | 416
  White | 465 | 480 | 945
  Other | 108 | 331 | 439
Professional Role [Count of Participants; unit: Participants]
  Clinician | 77 | 219 | 296
  Nurse | 305 | 540 | 845
  Assistant or Technician | 300 | 285 | 585
  Administrative or Other | 180 | 171 | 351
Time at Site [Count of Participants; unit: Participants]
  <= 5 years | 535 | 696 | 1231
  >5 years | 327 | 519 | 846
Time in Profession [Count of Participants; unit: Participants]
  <= 5 years | 348 | 419 | 767
  > 5 years | 514 | 796 | 1310

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity
Description: Posttraumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual (DSM) of Mental Disorders (PCL-5). The PCL-5 is a 20-item measure of PTSD symptom severity. Each item is rated on 0-4 frequency scale. Items are summed to create a total score ranging from 0-80 where a higher score indicates worse outcomes.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 845 | 1192
score on a scale
  pre-intervention | 16.36 (15.87) | 17.10 (16.59)
  post-intervention | 15.56 (16.00) | 15.78 (16.17)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .77, Mixed Models Analysis; Mean Difference (Net) = 0.189, 95% CI 2-sided [-1.068 to 1.446] — Effect sizes are the difference between SFA minus Usual Care

2. Primary Outcome: Psychological Distress
Description: Kessler 6 Distress Scale (K-6) for general psychological distress in the past 30 days. This is a 6-item inventory. Each of the items is scored from "none of the time" (0) to "all of the time" (4). Items are summed for a total score ranging from 0-24 where a higher score indicates worse outcomes.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 857 | 1210
score on a scale
  pre-intervention | 5.56 (5.23) | 5.99 (5.47)
  post-intervention | 5.74 (5.51) | 5.74 (5.52)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .39, Mixed Models Analysis; Median Difference (Net) = 0.238, 95% CI 2-sided [-0.310 to 0.785] — Effect sizes are the difference between SFA minus Usual Care

3. Secondary Outcome: Sleep-Related Impairment
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment (SRI) includes 4 items to assess sleep impairment over the past seven days. Each of the items are rated from 1-5 (not at all to very much). Items are summed into a scale ranging from 4-20 where a higher score indicates worse outcomes.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 861 | 1211
score on a scale
  pre-intervention | 9.83 (4.61) | 9.65 (4.53)
  post-intervention | 9.53 (4.60) | 9.56 (4.50)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .24, Mixed Models Analysis; Mean Difference (Net) = -0.232, 95% CI 2-sided [-0.618 to 0.153] — Effect sizes are the difference between SFA minus Usual Care

4. Secondary Outcome: Workplace Stress
Description: American Psychological Association's (APA) Stress in the Workplace survey; 3 items rated on a 1-5 scale from strongly disagree to strongly agree. A summed scale is formed ranging from 3-15 in which a higher score indicates worse outcomes/more stress.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 860 | 1210
score on a scale
  pre-intervention | 7.43 (2.79) | 7.78 (2.90)
  post-intervention | 7.79 (2.73) | 7.98 (2.83)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .23, Mixed Models Analysis; Median Difference (Net) = 0.134, 95% CI 2-sided [-0.085 to 0.352] — Effect sizes are the difference between SFA minus Usual Care

5. Secondary Outcome: Resilience
Description: Connor Davidson Resilience Scale (CDRISC); a brief (2-item) version of the scale with items rated from 0-4 (not true at all to true nearly all the time). Items are summed into a total scale ranging from 0-8 in which a higher score indicates better outcomes.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 861 | 1211
score on a scale
  pre-intervention | 6.39 (1.35) | 6.27 (1.44)
  post-intervention | 6.31 (1.39) | 6.22 (1.44)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .44, Mixed Models Analysis; Median Difference (Net) = -0.051, 95% CI 2-sided [-0.179 to 0.078] — Effect sizes are the difference between SFA minus Usual Care

6. Secondary Outcome: Burnout
Description: Dolan single item with 5 responses options ranging from 1[I enjoy my work. I haven symptoms of burnout.] to 5 [I feel completely burned out.]; We created a binary indicator to measure the percent of participants who reported experiencing symptoms of burnout.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 770 | 1159
Participants
  pre-intervention | 377 | 570
  post-intervention | 393 | 589
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .85, Repeated measure logistic regression; using GEE method; Odds Ratio, log = -0.051, 95% CI 2-sided [-0.179 to 0.078] — Effect sizes are the difference between SFA minus Usual Care

7. Secondary Outcome: Moral Distress
Description: We used the Moral Distress Thermometer, a single item sliding scale with responses rated on a 0-10 scale (none to worst possible) where a higher score indicates worse outcomes.
Time Frame: Pre-Intervention (Baseline) and Post-Intervention (29 to 53 days from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stress First Aid | Usual Care
Number analyzed (Participants) | 854 | 1208
score on a scale
  pre-intervention | 2.82 (2.62) | 3.35 (2.85)
  post-intervention | 2.85 (2.79) | 3.17 (2.80)
Statistical Analysis 1: Comparison: Stress First Aid vs Usual Care; Test type: Other — Standard 2-sided non-equivalence test; p = .08, Mixed Models Analysis; Median Difference (Net) = 0.230, 95% CI 2-sided [-0.025 to 0.484] — Effect sizes are the difference between SFA minus Usual Care

ADVERSE EVENTS:
Description: This trial included health professionals as participants and the intervention was low to no risk because it was a prevention approach. We did not monitor any adverse events because participation involved completing Web-based surveys by self-report. Thus, the research team had no direct interaction with participants so there would be no way to know of any adverse events.
Arm/Group | Stress First Aid | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Response rate was low (only 28% completed both the pre-intervention and post-intervention surveys).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04723576/Prot_SAP_000.pdf